CLINICAL TRIAL: NCT06557629
Title: Reaching a Caloric Goal Using a Gastric Sonar Versus Aspiration of Gastric Contents in Critically Ill Patients Receiving Nasogastric Enteral Nutrition - Randomized Controlled Trial
Brief Title: Reaching a Caloric Goal Using a Gastric Sonar Versus Aspiration of Gastric Contents in Critically Ill Patients Receiving Nasogastric Enteral Nutrition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0177-24-MMC
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Enteral Nutrition Intolerance in Critically Ill Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): Assessment of gastric residual volume via US
  Interventions: Diagnostic Test: Ultrasound assessment
- Aspiration group (No Intervention): assessment of gastric residual volume via aspiration of gastric content

INTERVENTIONS:
Diagnostic Test: Ultrasound assessment — Ultrasound assessment of gastric residual volume
  Arms: Ultrasound group

SUMMARY:
Enteral nutrition intolerance, manifested in delayed gastric emptying and high gastric residual, is a common problem in critically ill patients in intensive care, with adverse consequences on patients' outcomes. A decrease in the levels of the ghrelin hormone in these patients may contribute to this problem. The gastric residual test (GRV) is used to assess enteral absorption and gastric motility, but the traditional methods can lead to inaccuracy and waste of resources. In recent years, the use of ultrasound (PoCUS) to assess GRV has developed, but its effect on the rate of reaching the caloric goal has not yet been evaluated.

ELIGIBILITY:
Inclusion Criteria: Adult intensive care patients who recieve enteral nutrition via nasogastric tube -

Exclusion Criteria: 1. Pregnant patient 2. History of bariatric or other gastric surgery 3. Post-operative patients with sub-costal incision 4. Diaphragmatic hernia 5. Patients who recieve parenteral nutrition 6. Technically difficult US exam

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Reaching the daily caloric goal | 3 days
  To compare the daily caloric goal via gastric residual volume assessment with ultrasound vs. gastric aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel